CLINICAL TRIAL: NCT06446804
Title: Feedback on the Use of Eptinezumab: Efficacy at 6 Months in Severe Migraine
Brief Title: Follow-up of Migraine Patients on Eptinezumab
Acronym: EPTI-CO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2024/AL-01
Record Dates: First submitted 2024-05-30; First posted 2024-06-06 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Migraine patients: Patients with severe migraine, with at least 8 migraine days per month and at least 2 failed background treatments.
  Interventions: Other: None, pure observationnal study

INTERVENTIONS:
Other: None, pure observationnal study — Pure observatonnal study

SUMMARY:
The October 2022 Transparency Commission considers that VYEPTI (eptinezumab) is a treatment option for patients suffering from severe migraine with at least 8 migraine days per month, who have failed at least two prophylactic treatments and have no cardiovascular impairment.

Since the beginning of 2023, eptinezumab has been available in France as an inpatient treatment prescribed by a migraine neurologist in a growing number of centres. The Saint-Denis Hospital and the Nîmes University Hospital are among the first centres to have started. The investigators from these 2 centres have therefore decided to pool their data to provide the first French feedback on its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients suffering from severe migraine with at least 8 migraine days per month

  * Patients who have failed at least 2 disease-modifying treatments,
  * Patients treated with quarterly infusions of eptinezumab since March 2023 in a day hospital at Saint-Denis Hospital and Nîmes University Hospital.

Exclusion Criteria:

* Patient refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with severe migraine with at least 8 migraine days per month and failure of at least 2 disease-modifying therapies, treated with quarterly infusions of eptinezumab since March 2023 in a day hospital at the Saint-Denis hospital and the Nîmes university hospital.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Headaches and migraines per month | 6 months
  Number of headache and migraine days per month.
Responders | 6 months
  Rate of responders (30%, 50% and super responders > 75%)
Duration | 6 months
  Duration of effect of eptinezumab infusion (Numbers of weeks)
HIT6 scores (disability score) | 6 months
  Evaluation of HIT6 scores (disability score),
  ≤ 49 headaches have little impact on daily life; between 50 and 55: headaches have some impact on daily life; 56 to 59: headaches have a significant impact on daily life; ≥ 60
HAD (anxiety/depression score) | 6 months
  Evaluation of HAD score. From 0 to 7: absence of anxiety and/or depressive disorders, from 8 to 10: doubtful symptomatology, 11 to 21: proven anxiety and/or depression disorders of varying severity.
Concomitant treatments | 6 months
  Use of concomitant crisis and background treatments (description)

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (2):
- France (2):
  - CHU de Nîmes, Nîmes
  - CH de Saint Denis, Saint-Denis